CLINICAL TRIAL: NCT04666324
Title: Effects of Simethicone and Multilac Baby on Fecal Calprotectin Levels Infantile Colic
Brief Title: Effects of Multilac Baby on Fecal Calprotectin Levels of Colicky Babies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kalisz 2020-02
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simethicone Solution (Active Comparator): Treatment with simethicone (Espumisan®, 100 mg/ml, Berlin-Chemie / Menarini Polska Sp z o.o., Warsaw, Poland) for four weeks. Simethicone was administered 3-6 times per day with each treatment comprising 6 drops of the 100 mg/ml emulsion.
  Interventions: Drug: Simethicone Solution
- Multilac Baby (Experimental): Treatment with one stick pack of the multi-strain synbiotic (Multilac® Baby, Vivatrex GmbH, Aachen, Germany) per day for four weeks. Each stick pack of Multilac® Baby contains a total of 10^9 colony forming units (CFU) with equal CFU amounts of the following probiotic bacteria: L. acidophilus LA-14, L. casei R0215; L. paracasei Lpc-3; L. plantarum Lp-115; L. rhamnosus GG, L. salivarius Ls-33, B. lactis Bl-04, B. bifidum R0071, B. longum R0175 and 1.43 g of the prebiotic fructooligosaccharides.
  Interventions: Dietary Supplement: Multilac Baby

INTERVENTIONS:
Drug: Simethicone Solution — Oral daily treatment for four weeks
  Other Names: Control Group
  Arms: Simethicone Solution
Dietary Supplement: Multilac Baby — Oral daily treatment for four weeks
  Other Names: Treatment Group
  Arms: Multilac Baby

SUMMARY:
Open trial with two parallel arms, assessing the effects of Simethicone and Multilac Baby on crying behavior and fecal calprotectin levels in babies diagnosed for infantile colic.

DETAILED DESCRIPTION:
Babies aged 3 to 6 weeks will be diagnosed for infantile colic using the Wessel's criteria. Study design will be open label with two parallel arms (Simethicone and Multilac Baby). Multilac Baby is a synbiotic product containing probiotic bacteria (six lactobacilli and 3 bifidobacteria). Effects of treatments on crying behavior will be assessed by using parental 24h paper diaries. Fecal calprotectin values at the beginning and at the end of the study will be evaluated using BÜHLMANN Quantum Blue® Calprotectin High Range (Schönenbuch, Switzerland), a quantitative immunoassay.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed for infantile colic according to Wessel's criteria

Exclusion Criteria:

* previous treatment with probiotic or synbiotic
* previous treatment with antibiotics

Ages: 3 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change of days of crying | Three weeks
  Measurement of days of crying during last three weeks before enrollment and before the end of treatment. Treatment success will be determined by calculation the percentage of patients for whom the measurement will be reduced by the respective treatment by equal or more than 50 percent, compared to the value at the time of enrollment.
Change of average duration of evening crying | Three weeks
  Measurement of average duration of evening crying during last three weeks before enrollment and before the end of treatment. Treatment success will be determined by calculation the percentage of patients for whom the measurement will be reduced by the respective treatment by equal or more than 50 percent, compared to the value at the time of enrollment.
Change of fecal calprotectin values | 1-30 days
  BÜHLMANN Quantum Blue® Calprotectin High Range (Schönenbuch, Switzerland). It is a quantitative determination of fecal calprotectin through a sandwich immunoassay. Treatment success will be determined by calculation the percentage of patients for whom the measurement will be reduced by the respective treatment by equal or more than 50 percent, compared to the value at the time of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Krauss, Prof., Principal Investigator — The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz
Locations (2):
- Poland (2):
  - GP Clinic "Panaceum", Brody
  - GP Clinic "Pro Familia", Koziegłowy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Piatek J, Krauss H, Ciechelska-Rybarczyk A, Bernatek M, Wojtyla-Buciora P, Sommermeyer H. In-Vitro Growth Inhibition of Bacterial Pathogens by Probiotics and a Synbiotic: Product Composition Matters. Int J Environ Res Public Health. 2020 May 11;17(9):3332. doi: 10.3390/ijerph17093332. PMID 32403297
- [Derived] Sommermeyer H, Bernatek M, Pszczola M, Krauss H, Piatek J. Supporting the diagnosis of infantile colic by a point of care measurement of fecal calprotectin. Front Pediatr. 2022 Sep 29;10:978545. doi: 10.3389/fped.2022.978545. eCollection 2022. PMID 36245729
- [Derived] Bernatek M, Piatek J, Pszczola M, Krauss H, Antczak J, Maciukajc P, Sommermeyer H. Nine-Strain Bacterial Synbiotic Improves Crying and Lowers Fecal Calprotectin in Colicky Babies-An Open-Label Randomized Study. Microorganisms. 2022 Feb 12;10(2):430. doi: 10.3390/microorganisms10020430. PMID 35208884
- See also: Publication — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7246756/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT04666324/Prot_SAP_000.pdf